CLINICAL TRIAL: NCT01548573
Title: Tandem Autotransplantation for Multiple Myeloma in Participants With Less Than 12 Months of Preceding Therapy, Incorporating Velcade (Bortezomib) With the Transplant Chemotherapy and During Maintenance
Brief Title: Tandem Auto Transplantation in Myeloma Patients With <12 Months of Prior Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Met study stopping rules
Sponsor: University of Iowa (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Guido Tricot, Director, Holden Cancer Center Bone Marrow Transplant and Myeloma Program, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201202818; 7R01CA115399 (NIH)
Record Dates: First submitted 2012-02-29; First posted 2012-03-08 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; POEMS (Polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes); amyloidosis; bone marrow transplant; autologous
MeSH Terms: conditions — Multiple Myeloma; Polyneuropathies; Endocrine System Diseases; Paraproteinemias; Amyloidosis | interventions — Dexamethasone; Calcium Dobesilate; Cisplatin; Doxorubicin; Cyclophosphamide; Etoposide; Bortezomib; Thalidomide; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tandem autologous stem cell transplant (Experimental): Induction: DPACE(dexamethasone,cisplatin,doxorubicin,cyclophosphamide,etoposide) chemotherapy plus stem cell collection. Additional stem cell collection and/or chemotherapy may be required.
  After collection, participants will receive dexamethasone x 4 days every 14 days.
  Transplant 1: The transplant preparative regimen will be bortezomib/thalidomide/dexamethasone/melphalan.
  Once recovered, participants start thalidomide daily and dexamethasone x 4 days every 21 days.
  Consolidation (if administered): VDT-PACE(bortezomib,dexamethasone,thalidomide,cisplatin,doxorubicin,cyclophosphamide, etoposide) Transplant 2: 8 weeks to 6 months after the first transplant, participants will have the second transplant Maintenance: Year 1- VTD (bortezomib, thalidomide, dexamethasone) cycles. Year 2 - VCD (bortezomib, cyclophosphamide, dexamethasone)cycles.
  Interventions: Drug: Dexamethasone; Procedure: Tandem autologous stem cell transplant; Drug: Cisplatin; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Bortezomib; Drug: Thalidomide; Drug: Melphalan

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Procedure: Tandem autologous stem cell transplant
Drug: Cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: Doxorubicin — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: Cyclophosphamide — Given IV or PO
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: Etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213; Vepesid
Drug: Bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Drug: Thalidomide — Given PO
  Other Names: Kevadon; Synovir; THAL; Thalomid
Drug: Melphalan — Given IV
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin

SUMMARY:
This study is designed to decrease toxicity associated with prior tandem transplant protocols by reducing the intensity of induction, consolidation and maintenance therapy, while increasing event-free survival by adding bortezomib (Velcade®), thalidomide, gemcitabine and carmustine to the transplant regimens to down-regulate the rescue of myeloma cells by the micro-environment and to prevent DNA repair post high-dose alkylating agent therapy. By reducing drug resistance, it is hoped that 3-year event-free survival will be increased significantly when compared to Total Therapy II. Additionally, participants will have the option of providing biospecimens for a sub-study evaluating gene expression profiling at specific timepoints to better understand drug-resistance in myeloma, and to determine whether there are genes or gene products in the resistant population that can be targeted by novel therapies.

DETAILED DESCRIPTION:
This study is targeted towards patients who have been diagnosed with Multiple Myeloma, POEMS(Polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes), or myeloma plus amyloidosis and have had no more than 12 months of prior treatment. Furthermore, participants cannot have had a prior autologous or allogeneic transplant. The study schema consists of one round of induction chemotherapy, two transplants, one round of consolidation chemotherapy, and two years of maintenance treatment. This study design differs from its historical predecessors in the following manner:

* In contrast to Total Therapy II and III, which only allow enrollment of patients with one cycle or one month of treatment prior to enrollment, the proposed study allows enrollment of participants with up to 12 months of prior treatment.
* Induction therapy has been reduced to a single cycle.
* Bortezomib and thalidomide have been added to the transplant regimen.
* Carmustine is added to the second transplant.
* Gemcitabine is added to the second transplant regimen.
* Consolidation treatment has been reduced to a single cycle.
* The first year of maintenance consists of 12 28-day cycles of bortezomib,dexamethasone, and either thalidomide, lenalidomide, or cyclophoshamide. The second year of maintenance therapy consists of lenalidomide and dexamethasone.
* The novel agents thalidomide and bortezomib are not introduced upfront, but only with transplantation, consolidation, and maintenance.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have had a diagnosis of symptomatic MM, MM + amyloidosis, or POEMS (osteosclerotic myeloma: Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal protein, Skin changes) requiring treatment. Participants with a previous history of smoldering myeloma will be eligible if there is evidence of progressive disease requiring chemotherapy. Note that study participants do not need to have active disease at the time of study entry, as participants may have received up to 12 months of prior chemotherapy, which might have induced a response.
2. Protein criteria must be present (quantifiable M-component of IgG, IgA, IgD, or IgE and/or urinary kappa or lambda light chain, Bence-Jones protein, or Free Kappa Light Chain or Free Lambda Light Chain) in order to evaluate response. Non-secretory participants are eligible provided the participant has > 20% plasmacytosis OR multiple (>3) focal plasmacytomas or focal lesions on MRI.
3. Participants must have received no more than 12 months of prior chemotherapy for this disease. Participants may have received prior radiotherapy provided approval has been obtained from the PI.
4. Participants must not have had a prior transplant.
5. Participants must be 18-80 years of age at the time of study entry.
6. Ejection fraction by ECHO or MUGA of ≥ 40% performed.
7. Participants must have adequate pulmonary function studies, > 50% of predicted on mechanical aspects (FEV1, FVC) and diffusion capacity (DLCO) > 50% of predicted (adjusted for hemoglobin). If the participant is unable to complete pulmonary function tests due to disease related pain or condition, a participant may still be enrolled provided that the PI or enrolling investigator documents that the participant is a transplant candidate.
8. Participants must have a creatinine < 3 mg/dl and a calculated creatinine clearance >30mL/min. The Cockroft-Gault equation may be used to obtain calculated creatinine clearance.
9. Participants must have a performance status of 0-2 based on ECOG criteria. Participants with a poor performance status (3-4)based solely on bone pain will be eligible, provided there is documentation to verify this.
10. Participants must sign the most current IRB-approved study ICF (Informed Consent Form).

Exclusion Criteria:

1. Prior autologous or allogeneic transplant.
2. Platelet count < 30 x 109/L, unless myeloma-related. If MM-related, the enrolling investigator must document this.
3. > grade 3 neuropathy.
4. Known hypersensitivity to bortezomib, boron, or mannitol.
5. Uncontrolled diabetes.
6. Recent (< 6 months) myocardial infarction, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension, or difficult to control cardiac arrhythmias.
7. Participants must not have light chain deposition disease-related renal failure or creatinine >3 mg/dl.
8. Participants must not have a concurrent malignancy unless it can be adequately treated by surgical, non-chemotherapeutic intervention. Participants may have a history of prior malignancy, provided that he/she has not had any treatment within 365 days of study entry AND that life expectancy exceeds 5 years at the time of study entry.
9. Participants must not have life-threatening co-morbidities.
10. Women of child-bearing potential must have a documented negative pregnancy test documented within one week of study entry. Women and men of reproductive potential may not participate unless they have agreed, by signing the study ICF, to use effective contraceptive method(s) as outlined in that form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guido J Tricot, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tandem Transplant in MM <12 Mos of Prior Treatment: This was a single arm study for myeloma patients with <12 months of prior treatment to determine whether the incorporation of bortezomib into a tandem transplant regimen followed by 2 years of maintenance therapy would increase event-free survival.
Period: Overall Study
Arm/Group | Tandem Transplant in MM <12 Mos of Prior Treatment
Started | 19
Completed | 14
Not Completed | 5
Not completed — Death | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Tandem Transplant in MM <12 Mos of Prior Treatment
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants] — Population: Enrollment halted prematurely. Study met stopping rules. Outcomes will not be tracked and published
  Participants
    <=18 years | 0
    Between 18 and 65 years | 16
    >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] — Population: Enrollment halted prematurely. Study met stopping rules. Outcomes will not be tracked and published
  years | 59.4 [49 to 70.6]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Enrollment halted prematurely. Study met stopping rules. Outcomes will not be tracked and published.
  Participants
    Female | 8
    Male | 11
Region of Enrollment [Number; unit: participants] — Population: Enrollment halted prematurely. Study met stopping rules. Outcomes will not be tracked and published
  participants
    United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Event-Free Survival (EFS)
Description: To determine whether, in comparison to Total Therapy II, the median Event-Free Survival (EFS) can be increased from 4.8 years to 7.2 years, which represents an increase in median EFS of approximately 50%, based on an intent-to-treat analysis.
Time Frame: 8 years
Population: Enrollment halted prematurely. Study met stopping rules (3 or more of the first 20 participants died due to treatment-related toxicity).
  Data for outcome measure 1 were not collected.
Groups:
- Tandem Autologous Stem Cell Transplant: Induction and PBSC Collection:1 cycle of combination D-PACE (and peripheral blood stem cell collection. After collection, participants may receive interim dexamethasone at 20mg days 1-4 every 14 days.
  Transplant 1: 6 weeks after first day of D-PACE , but can occur as early as 4 weeks and as late as 6 months. Once recovered, participants start thalidomide daily and dexamethasone x 4 days every 21 days.
  Transplant 2: 8 weeks-6 months after the first transplant, participants will have second transplant. Once recovered, participants start thalidomide daily and dexamethasone x 4 days every 21 days.
  Consolidation Phase (if administered): 4 weeks-4 months after second transplant, participants may receive consolidation chemotherapy.
  Maintenance Phase year 1 and 2:The first year of maintenance will commence between 6 weeks-6 months after consolidation or 4 weeks-6 months after transplant if consolidation is skipped.
  DP
Arm/Group | Tandem Autologous Stem Cell Transplant
Number analyzed (Participants) | 0
Value | 0

2. Primary Outcome: Identification of Drug Resistant Genes
Description: To determine whether repeated bone marrow samples analyzed for gene expression profiling (GEP) can identify genes related to drug resistance in myeloma. The drug resistant genes or the gene products might then be targeted specifically to eradicate myeloma cells surviving tandem transplantation.
Time Frame: 5 years
Population: Enrollment halted prematurely. Study met stopping rules (3 or more of the first 20 participants died due to treatment-related toxicity).
  Data for outcome measure 2 were not collected.
Arm/Group | Tandem Transplant in MM <12 Mos of Prior Treatment
Number analyzed (Participants) | 0
Value | 0

3. Secondary Outcome: Number of Grade 3 Non-hematologic and Grade 4 Hematologic Serious Adverse Events Associated With the Addition of Bortezomib, Thalidomide, and Dexamethasone Into Autologous Transplant Regimens.
Description: To determine whether bortezomib, thalidomide and dexamethasone with transplant 1 and velcade/gemcitabine with transplant 2 can be safely incorporated into well-tested pre-transplant regimens of high-dose melphalan and carmustine/melphalan in doses equivalent to the BEAM(BCNU, etoposide, arabinoside, melphalan)regimen. Treatment-related toxicities will be compared to those reported in the literature using similar intensive approaches.
Time Frame: 2 years
Population: Enrollment halted prematurely. Study met stopping rules (3 or more of the first 20 participants died due to treatment-related toxicity).
  Data for outcome measure 3 were not collected.
Arm/Group | Tandem Transplant in MM <12 Mos of Prior Treatment
Number analyzed (Participants) | 0
Value | 0

4. Secondary Outcome: Overall Survival
Description: To determine the median overall survival based on an intent-to-treat analysis, which should exceed 10 years, based on the projected 10-year survival of Total Therapy III, keeping in mind that participants are included in this protocol with up to 12 months of prior therapy.
Time Frame: 10 years
Population: Enrollment halted prematurely. Study met stopping rules (3 or more of the first 20 participants died due to treatment-related toxicity).
  Data for outcome measure 4 were not collected.
Arm/Group | Tandem Transplant in MM <12 Mos of Prior Treatment
Number analyzed (Participants) | 0
Value | 0

ADVERSE EVENTS:
Arm/Group | Tandem Transplant in MM <12 Mos of Prior Treatment
All-Cause Mortality (participants affected / at risk) | 3/19
Serious Adverse Events (participants affected / at risk) | 13/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tandem Transplant in MM <12 Mos of Prior Treatment (N=19)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 1 (1)
Stoke secondary to cardio-embolism (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Fever (General disorders) | 2 (2)
Chest pain, air embolism (Cardiac disorders) | 1 (1)
Neutropenic fever (General disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fever (General disorders) | 3 (3)
Myocardial infarction (Cardiac disorders) | 1 (1)
Malaise and abrupt chest pain (General disorders) | 1 (1)
Neutropenic fever, abdominal pain, and loose stools (General disorders) | 1 (1)
Respiratory distress, fevers, and pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea, and abdominal pain (Gastrointestinal disorders) | 1 (1)
Nausea, failure-to-thrive, and line-associated deep vein thrombosis (Blood and lymphatic system disorders) | 1 (1)
Atrial Fibrillation with RVR (Cardiac disorders) | 2 (2)
Hypoxia, fever, pulmonary infiltrates with nodules, and C Diff + diarrhea (General disorders) | 1 (1)
Viral pneumonia (Infections and infestations) | 1 (1)
Chills, cough, throat pain, dyspnea. Mucositis. + hMPV. Engraftment syndrome (General disorders) | 1 (1)
Severe back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pneumonia, Atrial fib w/ cardioversion (Cardiac disorders) | 1 (1)
Acute kidney injury, uncontrolled hypertension, thrombotic microangiopathy (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tandem Transplant in MM <12 Mos of Prior Treatment (N=19)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Abdominal Pain/discomfort LLQ (Gastrointestinal disorders) | 1 (1)
Abdominal Pain/discomfort RUQ (Gastrointestinal disorders) | 1 (1)
Activated PTT prolonged (Investigations) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Akathisia (restless feet) (Nervous system disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4)
Allergic reaction during PBSC Collection (Investigations) | 1 (1)
ALT increased (Investigations) | 5 (6)
Anemia (Blood and lymphatic system disorders) | 19 (65)
Anemia (Hemolytic) (Blood and lymphatic system disorders) | 1 (1)
Ankle edema (General disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (8)
Anxiety (Psychiatric disorders) | 1 (2)
aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
AST increased (Investigations) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 2 (3)
Atrial Fibrillation with RVR (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Bilateral Calf Pain at time of engraftment (Musculoskeletal and connective tissue disorders) | 1 (1)
Bilateral edema in limbs (General disorders) | 1 (1)
Bleeding at port site (General disorders) | 1 (1)
Bleeding from hemorrhoids (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 3 (3)
Blurred vision (Eye disorders) | 2 (2)
Bone marrow hypocellularity (Blood and lymphatic system disorders) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone/joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Bruising on abdomen and arms (Injury, poisoning and procedural complications) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Catheter related infection: enterococcal (vanc sensitive) (Infections and infestations) | 2 (2)
Catheter-related infection (Infections and infestations) | 1 (1)
catheter-related infection (gram+ cocci) (Infections and infestations) | 1 (1)
Catheter-related infection (VRE) (Infections and infestations) | 1 (1)
Catheter-related infection: enterococcal (vanc sensitive) (Infections and infestations) | 1 (1)
C-Diff colitis (Gastrointestinal disorders) | 1 (1)
chest pain-cardiac (Cardiac disorders) | 1 (1)
Cholecystitis (w/ gallstone present) (Hepatobiliary disorders) | 1 (1)
CMV Reactivation (Infections and infestations) | 1 (1)
Coag neg staph bacteremia x 3 (Infections and infestations) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Colitis (C-Diff) (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 2 (4)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 10 (11)
Diarrhea (c diff pos) (Gastrointestinal disorders) | 3 (4)
Diarrhea (C Diff Neg) (Gastrointestinal disorders) | 8 (8)
Diarrhea (C Diff) (Gastrointestinal disorders) | 2 (3)
Diarrhea/loose stools (Gastrointestinal disorders) | 1 (1)
Dizziness (General disorders) | 8 (10)
Dizziness (orthostatic hypotension) (General disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dygeusia (abnormal taste) (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dysgeusia (altered taste) (Nervous system disorders) | 1 (1)
Dysnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Gastrointestinal disorders) | 8 (12)
Ear Pain (Ear and labyrinth disorders) | 1 (1)
Edema (General disorders) | 1 (1)
Edema (feet) (General disorders) | 1 (1)
Edema in left lower ankle (General disorders) | 1 (1)
Edema Limbs (General disorders) | 1 (1)
Edema limbs (bilateral) (General disorders) | 1 (1)
Edema limbs (legs) (General disorders) | 1 (1)
Engraftment fever (General disorders) | 1 (1)
Engraftment fevers (Blood and lymphatic system disorders) | 1 (1)
Engraftment fevers controlled with steroids (General disorders) | 1 (1)
Engraftment syndrome (Immune system disorders) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Esophagitis (CMV related) (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 13 (26)
Febrile Neutropenia (Blood and lymphatic system disorders) | 10 (10)
Fever (General disorders) | 1 (1)
Fever (non-neutropenic) (General disorders) | 5 (6)
Flushing (Vascular disorders) | 1 (1)
Gait Disturbance (General disorders) | 1 (1)
Gait disturbance (d/t dizziness) (General disorders) | 1 (1)
Gallbladder sludge (Hepatobiliary disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (2)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Gastro-esophageal reflux (Gastrointestinal disorders) | 2 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Generalized bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
GERD with Barrett's esophagus (Gastrointestinal disorders) | 1 (1)
Hallucinations (with voriconazole) (Psychiatric disorders) | 1 (1)
Hand tremor (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (7)
Headache with dexamethasone (Nervous system disorders) | 1 (1)
HHV 6 viremia reactivation (Infections and infestations) | 1 (1)
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (14)
Hyperglycemia (Dex) (Metabolism and nutrition disorders) | 9 (15)
Hyperhidrosis (excessive perspiration) (Skin and subcutaneous tissue disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 4 (4)
Hypertension (Vascular disorders) | 3 (5)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 18 (42)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 12 (22)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Musculoskeletal and connective tissue disorders) | 6 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 16 (31)
Hypotension (Vascular disorders) | 5 (5)
Hypotension with PBSC infusion (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Infusion Site Extravasation w bruising, no pain (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Insomnia (Dex) (Psychiatric disorders) | 5 (5)
Iron overload (Metabolism and nutrition disorders) | 1 (1)
Joint pain right knee (Musculoskeletal and connective tissue disorders) | 1 (1)
joint pains in right hip and shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Left hemiparesis (Nervous system disorders) | 1 (1)
Left Rib Fracture (Injury, poisoning and procedural complications) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Lip infection (HSV) (Infections and infestations) | 1 (1)
Localized edema (leg) (General disorders) | 1 (1)
Localized edema (right leg) w/out DVT (General disorders) | 1 (1)
Low back and hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Lung infection: fungal pneumonia (Infections and infestations) | 1 (1)
Lung infection: left lower lobe consolidation (Infections and infestations) | 1 (1)
Lung infection: pneumonia (Infections and infestations) | 2 (2)
Lung infection: pneumonia (hMPV and staph) (Infections and infestations) | 1 (1)
Lung infection: Pulmonary infiltrates with nodules (Infections and infestations) | 1 (1)
Lung infection: RSV Pneumonia (Infections and infestations) | 1 (1)
Lung Infection: serratia marcescens (Infections and infestations) | 1 (1)
Lung infection: viral pneumonia (Infections and infestations) | 1 (1)
Lung infections: CMV pneumonia (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 19 (31)
Lymphopenic fever (Infections and infestations) | 1 (1)
Maculopapular rash (Skin and subcutaneous tissue disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Minor left leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Mucositis (morphine prn) (Gastrointestinal disorders) | 1 (1)
Mucositis (oral) (Gastrointestinal disorders) | 1 (1)
Mucositis (oral) requiring TPN (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (7)
Mucositis oral (cvn + pca narcotics) (Gastrointestinal disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (24)
Nausea with dexamethasone (Gastrointestinal disorders) | 1 (1)
Nausea/vomiting (from post-nasal drip) (Gastrointestinal disorders) | 1 (1)
Nausea/Vomiting (TPN) (Gastrointestinal disorders) | 1 (1)
Neutropenic fever (General disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Non-cardiac pleuritic chest pain (General disorders) | 1 (1)
Oral pain (tongue lesion) (Gastrointestinal disorders) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 1 (1)
Other, muscle spasms in lower back and neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Other: Chloride increased (Metabolism and nutrition disorders) | 1 (1)
Other: CMV reactivation (Infections and infestations) | 1 (1)
Other: CO2 decreased (Metabolism and nutrition disorders) | 1 (1)
Other: Failure to thrive (General disorders) | 2 (2)
Other: Left carotid artery stenosis (Vascular disorders) | 1 (1)
Other: Platelet refractoriness (Blood and lymphatic system disorders) | 1 (1)
Other: sub-therapeutic INR (Investigations) | 1 (1)
Other: Vanc sensitive Enterococcal + coag neg staph bacteremia (Investigations) | 1 (1)
Other: VRE + coag neg staph bacteremia (Enterococcus faecium) (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain at port and catheter site (General disorders) | 1 (1)
Pain in both elbows (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (left lower arm) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in hips and left lower leg (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in lower back (Musculoskeletal and connective tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pansinusitis (Infections and infestations) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral Neuropathy (Nervous system disorders) | 4 (7)
Peripheral Neuropathy (feet) (Nervous system disorders) | 1 (2)
Peripheral neuropathy (hands) (Nervous system disorders) | 1 (1)
Peripheral Neuropathy (thal held) (Nervous system disorders) | 1 (1)
Peripheral Neuropathy (thalidomide stopped) (Nervous system disorders) | 1 (1)
Peripheral Neuropathy (toes) (Nervous system disorders) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 19 (65)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (hMPV) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Post-nasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PTT prolonged (Investigations) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Rash - face and neck (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Respiratory failure/ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rib pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Rt knee joint pain w/ swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Scalp Pain (Skin and subcutaneous tissue disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sepsis (Gram Neg) (Infections and infestations) | 1 (1)
Serum amylase increased (Investigations) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Somnolence (Nervous system disorders) | 3 (3)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Stomach pain (not during dex admin) (Gastrointestinal disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Swelling of right hand (neg doppler) (General disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Toe infection (Infections and infestations) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Tremor in hands, R> L (Nervous system disorders) | 2 (2)
Urinary Frequency (Renal and urinary disorders) | 1 (1)
Urinary Frequency (Nocturnal) (Renal and urinary disorders) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (3)
Vancomycin-Resistant Enterococcus (Infections and infestations) | 2 (2)
Vascular Access Complication (air embolism) (Injury, poisoning and procedural complications) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (9)
WBC decreased (Investigations) | 19 (56)
Weakness (General disorders) | 2 (4)
Weight Loss (Investigations) | 3 (4)

LIMITATIONS AND CAVEATS:
Enrollment halted prematurely. Study met stopping rules. Outcomes will not be tracked and published

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes